CLINICAL TRIAL: NCT06131385
Title: Registration of Intravenous Thrombolysis for Acute Ischemic Stroke in Southwestern China（IVTIS）
Acronym: IVTIS
Status: Recruiting | Type: Observational
Sponsor: Zhengzhou Yuan (Other)
Responsible Party: Sponsor-Investigator, Zhengzhou Yuan, Deputy Director of Stroke Center, The Affiliated Hospital Of Southwest Medical University
Organization: The Affiliated Hospital Of Southwest Medical University (Other)
Other Study IDs: SWMU-2023-12
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute ischemic stroke treated with intravenous thrombolysis: All of acute ischemic stroke patients who treated with intravenous thrombolysis.
  Interventions: Drug: intravenous thrombolysis

INTERVENTIONS:
Drug: intravenous thrombolysis — Intravenous thrombolysis using thrombolytic drugs such as ateplase and teneplase.

SUMMARY:
This study aims to observe the safety and effectiveness of intravenous thrombolysis for acute ischemic stroke in real-world clinical practice.

DETAILED DESCRIPTION:
IVTIS is a prospective, real-world registry lasting for 22 years. A total of 3000 patients with intravenous thrombolysis will be enrolled。

ELIGIBILITY:
Inclusion Criteria:

* The patient was diagnosed with acute ischemic stroke and received intravenous thrombolysis.

Exclusion Criteria:

* No additional exclusion criteria.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute ischemic stroke who received intravenous thrombolysis will be included in the study and no additional exclusion criteria have been set.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2045-12-15 (Estimated); Study Completion 2046-05-01 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) score | 90±7 days
  Ordinal distribution of mRS at 90±7 days; modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)

SECONDARY OUTCOMES:
Excellent functional outcome | 90±7 days
  Proportion of subjects with mRS 0-1 at 90±7 days.
Good functional outcome | 90±7 days
  Proportion of subjects with mRS 0-2 at 90±7 days.
mRS 0-3 | 90±7 days
  Proportion of subjects with mRS 0-3 at 90±7 days.
Change of National Institutes of Health Stroke Scale (NIHSS) | 24 hours
  Change of National Institutes of Health Stroke Scale (NIHSS, a scale between 0 and 42 on which higher scores indicate more severe neurologic deficits) from baseline to 24 hours.
Change of National Institutes of Health Stroke Scale (NIHSS) | 7 days
  Change of National Institutes of Health Stroke Scale (NIHSS, a scale between 0 and 42 on which higher scores indicate more severe neurologic deficits) from baseline to 7 days.
Symptom-to-thrombolysis time | 24 hours
  Time from onset of symptoms to thrombolytic therapy.
Door-to-Needle Time | 24 hours
  Time from the arrival of stroke patient in emergency to initiation of thrombolysis therapy.
Incidence of clinically significant intracranial hemorrhage | 36 hours
  Incidence of sICH (Heidelberg criteria) measured at 36 hours
Incidence of any intracranial hemorrhage | 36 hours
  Incidence of any intracranial hemorrhage (Heidelberg criteria) measured at 36 hours
All-cause mortality | 90±7 days
  All-cause mortality at 90±7 days
Complications related to intravenous thrombolysis | up to 7 days
  Complications related to intravenous thrombolysis during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Zhengzhou Yuan, Study Chair — Department of Neurology, Affiliated Hospital of Southwest Medical University, Lu
Locations (1):
- Affiliated Hospital of Southwest Medical University, Luzhou, China

IPD SHARING:
Plan to Share IPD: Undecided